CLINICAL TRIAL: NCT03583190
Title: Comparing the Use of Cervical-Cranial Dry Needling With Orthopedic Manual Therapy to the Cervical Spine for Cervicogenic Headache: A Multi-center RCT With 1-Year Follow Up
Brief Title: Cervical-Cranial Dry Needling vs. Orthopedic Manual Therapy for Cervicogenic Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Youngstown State University (Other)
Collaborators: Franklin Pierce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0177-08
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cervicogenic Headache
Keywords: Neck pain; Headache; Dry needling; manual therapy
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain; Headache | interventions — Exercise; Patient Education as Topic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The outcome assessor will be blinded the treatment group. The clinician providing treatment will be blinded to outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical-cranial dry needling (Experimental): Patients randomized to this arm will receive cervical-cranial dry needling, thoracic manipulation, and exercise.
  Interventions: Other: Cervical-cranial dry needling; Other: Thoracic Manipulation; Other: Exercise; Other: Patient Education
- Orthopedic Manual Therapy (Active Comparator): Patients randomized to this arm will receive orthopedic manual therapy to cervical spine, thoracic manipulation, and exercise.
  Interventions: Other: Orthopedic manual therapy; Other: Thoracic Manipulation; Other: Exercise; Other: Patient Education

INTERVENTIONS:
Other: Cervical-cranial dry needling — Segmental needling of the neck and needling in the patient's headache distribution. Peripherally sensitized areas of the neck may also be dry needled based on the findings of the clinical evaluation.
  Arms: Cervical-cranial dry needling
Other: Orthopedic manual therapy — Orthopedic Manual Therapy (OMT) that includes either mobilization or manipulation to the cervical spine applied pragmatically to the most symptomatic level.
  Arms: Orthopedic Manual Therapy
Other: Thoracic Manipulation — Thoracic Manipulation (applied pragmatically) to the levels determined to be provocative or hypomobile.
Other: Exercise — Clinicians select 1 active range of motion exercise for the cervical spine, deep cervical flexion endurance exercise, and 5 upper extremity exercises (from a set of 10). Additionally, patients will be assigned a headache management technique.
Other: Patient Education — Patients will receive education regarding their headache condition, proper performance of their symptom management technique, posture.

SUMMARY:
Dry needling is a therapeutic modality used to treat a number of neuromusculoskeletal conditions. Practice trends suggest it is becoming widely used by Physical Therapists to help patients manage symptoms associated with CGH, however, there is limited scientific evidence demonstrating meaningful impact for dry needling for CGH. Manual therapy (thrust and non-thrust mobilizations) to the cervical spine are well researched and have an established treatment effect for managing symptoms related to CGH. The purpose of this study is to compare outcomes (1 week, 1 month, 3 months, 12 months) for patients with CGH treated with cervical-cranial dry needling or pragmatically applied orthopedic manual therapy to the cervical spine. In addition to either the cervical-cranial dry needling or manual therapy to the cervical spine, patients will also receive patient education, thoracic manipulation, and exercise.

DETAILED DESCRIPTION:
The use of dry needling is becoming widely used by Physical Therapists in the United States for a number of neuromusculoskeletal conditions including cervicogenic headache (CGH). Dry needling is performed by taking a mono-filament needle and inserting it into symptomatic soft tissue. In this trial, the dry needling will be performed segmentally in the neck and along the patient's headache distribution pattern. Orthopedic manual therapy (OMT) may include both thrust and non-thrust techniques applied to a targeted spinal level and has a well-established treatment effect for patients with CGH. In this trial, the OMT will be applied pragmatically to the cervical spine at the most symptomatic level of the headache. Other interventions used in this trial will include patient education, thoracic manipulation and exercise.

Patients will be randomized to receive either dry needling or OMT 2x/week for 2 weeks and then 1-2x/week for 2 weeks totaling 6-8 visits over the course of 1 month. The 1 week and 1 month outcomes collected will be reported on separately from the 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Meets the IHS criteria for CGH
* Headache frequency of at least 1 per week over a period greater than 3 months.
* Demonstrates segmental dysfunction with passive mobility testing.

Exclusion Criteria:

Patients whose headache experience is primarily of migraine origin. Tension-type headache, headache pain <2, contraindications to the interventions (malignancy, myelopathy, fracture, metabolic disease, rheumatoid arthritis, long-term corticosteroid use), headache presentation suggesting cervical arterial insufficiency, severe metal allergy, needle phobia, history of neck or thoracic spine surgery, Non-English speaking patients, therapist is unable to elicit the headache with passive accessory intervertebral movements (PAIVM), or pending litigation for neck pain and/or headache.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in NPRS headache intensity | Baseline, 1 week, 1 month, 3 months, 12 months.
  Average and most intense in the last week will be recorded using a 0 (no headache) to 10 (most intense)

SECONDARY OUTCOMES:
Change in disability using Neck Disability Index | Baseline 1 week, 1 month, 3 months, 12 months
  The NDI is a self-report measure of perceived disability comprised of ten questions using an ordinal scale from 0 to 5 for a maximum of 50 points.
Change in disability using Headache Disability Index (HDI) | Baseline, 1 week, 1 month, 3 months, 12 months
  The HDI assesses "the burden of chronic headaches," using 25 items that ask about the perceived impact of headaches on emotional functioning and daily activities. Items were designed specifically to assess the concerns of individuals with recurrent headache disorders.
Leeds Assessment of Neuropathic Signs and Symptoms (LANSS) | Baseline
  Subjects identifying particular qualities about their pain (yes/no) that could suggest problems with how the nervous system is interpreting pain. There is a physical screening procedure involving a discriminate evaluation of different sensations (light touch, and sharp/dull) in an area of the subject's body (arm or leg) without pain compared to an area of their pain (neck or head). The questions and results from the physical testing are scored which can range from 0-24.
Change in Medication intake | Baseline, 1 week, 1 month, 3 months, 12 months
  Patients will identify the medications + dosage they have consumed to treat their headache in the past week.
Patient Satisfaction | 1 month
  Patient satisfaction will be assessed using the Patient Satisfaction Instrument (PSI) that measures several constructs related to clinical outcomes and patient care. The PSI consists of 12 questions rated using a scale, 1 (strongly disagree) to 5 (strongly agree).
Health care utilization | 3 and 12 months
  Healthcare utilization will be reported by subjects identifying on a form any provider they have seen for care of their headaches, treatments they have received, and cost for their headaches.
SANE Percent Recovery | 1 month
  Percent recovery will be measured using a global percentage of improvement is a measure of the patient's perception of the change in their condition.
Change in current NPRS neck or headache intensity | Baseline and Immediately post intervention
  Current level of headache or neck pain on a scale ranging from 0 (no headache) to 10 (most intense)

CONTACTS AND LOCATIONS:
Overall Officials: David Griswold, PhD, Principal Investigator — Associate Professor at Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sedighi A, Nakhostin Ansari N, Naghdi S. Comparison of acute effects of superficial and deep dry needling into trigger points of suboccipital and upper trapezius muscles in patients with cervicogenic headache. J Bodyw Mov Ther. 2017 Oct;21(4):810-814. doi: 10.1016/j.jbmt.2017.01.002. Epub 2017 Jan 6. PMID 29037632
- [Background] France S, Bown J, Nowosilskyj M, Mott M, Rand S, Walters J. Evidence for the use of dry needling and physiotherapy in the management of cervicogenic or tension-type headache: a systematic review. Cephalalgia. 2014 Oct;34(12):994-1003. doi: 10.1177/0333102414523847. Epub 2014 Mar 12. PMID 24623124
- [Background] Bond BM, Kinslow C. Improvement in clinical outcomes after dry needling in a patient with occipital neuralgia. J Can Chiropr Assoc. 2015 Jun;59(2):101-10. PMID 26136602